CLINICAL TRIAL: NCT03659851
Title: Pretreatment With Levosimendan In Patients Undergoing Left Ventricular Assist Device Implantation
Brief Title: Levosimendan In Patients Undergoing LVAD Implantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Nikola Bradic, MD, Principal Investigator, University Hospital Dubrava
Other Study IDs: UH Dubrava
Record Dates: First submitted 2018-06-24; First posted 2018-09-06 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2019-10

CONDITIONS: Left Ventricular Dysfunction; Right Ventricular Dysfunction; Biventricular Failure
Keywords: Heart failure; Left ventricular dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left; Ventricular Dysfunction, Right; Heart Failure | interventions — Simendan

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Levosimendan before LVAD implantation: Levosimendan use 24 hrs. before LVAD implantation
  Interventions: Drug: Levosimendan 2.5 MG/ML Injectable Solution
- Dobutamine/milrinone before LVAD implantation: Dobutamine/milrinone use 24 hrs. before LVAD implantation

INTERVENTIONS:
Drug: Levosimendan 2.5 MG/ML Injectable Solution — LVAD implantation
  Other Names: Simdax
  Groups: Levosimendan before LVAD implantation

SUMMARY:
According to the results from the literature, it has been shown that levosimendan usage 24-48 hours before LVAD implementation can improve short and long-term outcome in these patients regarding to the patients without preoperative pretreatment. The aim is to compare short and long-term outcome in patients who underwent to LVAD implementation and pretreated with levosimendan regarding the patient without pretreatment or with other medications.

DETAILED DESCRIPTION:
Left ventricular assist device (LVAD) implantation is accepted for treatment of end-stage heart failure, in both as the bridging to heart transplantation or as the destination therapy. These patients have highly impaired systolic function which contributes to global heart dysfunction. The main complication is arising of pulmonary vascular pressures and pulmonary vascular resistance (PVR) and, consequently, right heart dysfunction. From the data in literature, RV dysfunction exist in approximately 25%-40% of patients with implanted LVAD, and in approximately 20%-30% of those died or have need for the RV assist device due to RV failure refractory to medications. Capability of the RV to maintain appropriate output and the fill of the LVAD is the main point for correct LVAD functioning and patients' early and late postoperative outcome. Preimplantation evaluation by echocardiography estimation of RV function, geometry and tricuspid valve function are the criteria for the diagnose of RV dysfunction. Laboratory analysis which can lead to the diagnose of RV dysfunction are also included in preimplantation evaluation. Specific inotropic therapy in patients with moderate or severe RV dysfunction and/or dilatation can improve RV function in preimplantation period. This is predominantly important in patients who were on the prolonged inotropic support with beta-agonist therapy before LVAD implantation and in whom their beta receptors are exhausted. The investigators will exam the hemodynamic effects of levosimendan administrated day before in patients underwent LVAD implantation. Further, investigators will analyze and evaluate early and late outcome in participants with implanted LVAD.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for LVAD implantation

Exclusion Criteria:

* Known patient's allergy on medication
* Patient's disagreement for the procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In study will be observed all patients scheduled for LVAD implantation because of severe heart failure in which heart transplantation cannot be performed due to medical conditions. Further, in study will be observed all patients scheduled for LVAD implantation because of severe heart failure in which any other conservative/surgery therapy did not give positive results.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-06-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of laboratory parameters in patients who underwent LVAD implantation and pretreated with levosimendan or other inotropic day before surgery | 9 years
  Patients will be divided into two groups depending of administrated inotropic pretreatment (levosimendan or other inotropic medications) in preoperative period. Further, laboratory data will be collected and analyzed three times in day before surgery and every four hours during first postoperative day after LVAD implantation to estimate changes and improvement/worsening of laboratory parameters depending of preoperative treatment.
Measurement of hemodynamic parameters in patients who underwent LVAD implantation and pretreated with levosimendan or other inotrope day before surgery | 9 years
  Patients will be divided into two groups depending of administrated inotropic pretreatment (levosimendan or other inotropic medications) in preoperative period. Further, hemodynamic data will be collected and analyzed three times in day before surgery and every four hours during first postoperative day after LVAD implantation to estimate changes in hemodynamic outcome depending of preoperative treatment. Hemodynamic parameter 1 and its changes is systemic vascular resistance index (SVRI); expressed by dyn·sec/cm5/m2
Measurement of hemodynamic parameters in patients who underwent LVAD implantation and pretreated with levosimendan or other inotrope day before surgery | 9 years
  Patients will be divided into two groups depending of administrated inotropic pretreatment (levosimendan or other inotropic medications) in preoperative period. Further, hemodynamic data will be collected and analyzed three times in day before surgery and every four hours during first postoperative day after LVAD implantation to estimate changes in hemodynamic outcome depending of preoperative treatment. Hemodynamic parameter 2 and its changes is pulmonary vascular resistance index (PVRI), expressed by dyn·sec/cm5/m2
Measurement of hemodynamic parameters in patients who underwent LVAD implantation and pretreated with levosimendan or other inotrope day before surgery | 9 years
  Patients will be divided into two groups depending of administrated inotropic pretreatment (levosimendan or other inotropic medications) in preoperative period. Further, hemodynamic data will be collected and analyzed three times in day before surgery and every four hours during first postoperative day after LVAD implantation to estimate changes in hemodynamic outcome depending of preoperative treatment. Hemodynamic parameter 3 and its changes is cardiac index (CI) expressed by L/min per m2
Measurement of hemodynamic parameters in patients who underwent LVAD implantation and pretreated with levosimendan or other inotrope day before surgery | 9 years
  Patients will be divided into two groups depending of administrated inotropic pretreatment (levosimendan or other inotropic medications) in preoperative period. Further, hemodynamic data will be collected and analyzed three times in day before surgery and every four hours during first postoperative day after LVAD implantation to estimate changes in hemodynamic outcome depending of preoperative treatment. Hemodynamic parameter 4 and its changes is right stroke work indexes (RVSWI) expressed by g·m/m2/beat
Measurement of hemodynamic parameters in patients who underwent LVAD implantation and pretreated with levosimendan or other inotrope day before surgery | 9 years
  Patients will be divided into two groups depending of administrated inotropic pretreatment (levosimendan or other inotropic medications) in preoperative period. Further, hemodynamic data will be collected and analyzed three times in day before surgery and every four hours during first postoperative day after LVAD implantation to estimate changes in hemodynamic outcome depending of preoperative treatment. Hemodynamic parameter 5 and its changes is left stroke work indexes (LVSWI) expressed by g·m/m2/beat
Measurement of hemodynamic parameters in patients who underwent LVAD implantation and pretreated with levosimendan or other inotrope day before surgery | 9 years
  Patients will be divided into two groups depending of administrated inotropic pretreatment (levosimendan or other inotropic medications) in preoperative period. Further, hemodynamic data will be collected and analyzed three times in day before surgery and every four hours during first postoperative day after LVAD implantation to estimate changes in hemodynamic outcome depending of preoperative treatment. Hemodynamic parameter 6 and its changes is stroke volume index (SVI) expressed by mL/m2
Measurement of hemodynamic parameters in patients who underwent LVAD implantation and pretreated with levosimendan or other inotrope day before surgery | 9 years
  Patients will be divided into two groups depending of administrated inotropic pretreatment (levosimendan or other inotropic medications) in preoperative period. Further, hemodynamic data will be collected and analyzed three times in day before surgery and every four hours during first postoperative day after LVAD implantation to estimate changes in hemodynamic outcome depending of preoperative treatment. Hemodynamic parameter 7 and its changes is right ventricular end-diastolic volume (RVEDV) expressed by mL.
Measurement of echocardiography parameters in patients who underwent LVAD implantation and pretreated with levosimendan or other inotropic day before surgery | 9 years
  Patients will be divided into two groups depending of administrated inotropic pretreatment (levosimendan or other inotropic medications) in preoperative period. Echocardiography data will be collected and analyzed three times in day before surgery and every four hours during first postoperative day after LVAD implantation to estimate changes and improvement/worsening of echocardiography parameters depending of preoperative treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Nikola Bradic, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sponga S, Ivanitskaia E, Potapov E, Krabatsch T, Hetzer R, Lehmkuhl H. Preoperative treatment with levosimendan in candidates for mechanical circulatory support. ASAIO J. 2012 Jan-Feb;58(1):6-11. doi: 10.1097/MAT.0b013e318239f401. PMID 22157071
- [Background] Theiss HD, Grabmaier U, Kreissl N, Hagl C, Steinbeck G, Sodian R, Franz WM, Kaczmarek I. Preconditioning with levosimendan before implantation of left ventricular assist devices. Artif Organs. 2014 Mar;38(3):231-4. doi: 10.1111/aor.12150. Epub 2013 Oct 22. PMID 24147881